CLINICAL TRIAL: NCT05189366
Title: Sophrology Treatment for Patients With Glial Tumours Requiring Speech Therapy
Acronym: SOPHNEURO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ICO-2020-12
Record Dates: First submitted 2021-12-28; First posted 2022-01-12 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Glial Tumor
Keywords: Sophrology; Speech therapy
MeSH Terms: conditions — Glioma; Communication Disorders | interventions — Speech Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm : Speech therapy + Sophrology (Experimental): In the experimental arm, patients will receive 6 sessions of sophrology. The sessions are individual and last approximately 50 minutes.
  In addition to the sophrology sessions, patients will benefit from two speech therapy sessions per week for 6 months, lasting from 30 minutes to 1 hour depending on the patient's general condition.
  Interventions: Behavioral: Sophrology; Behavioral: Speech therapy
- Control arm : Speech therapy (Active Comparator): Patients will benefit from two speech therapy sessions per week for 6 months, lasting from 30 minutes to 1 hour depending on the patient's general condition.
  Interventions: Behavioral: Speech therapy

INTERVENTIONS:
Behavioral: Sophrology — Sophrology is a relaxation method that's sometimes referred to as hypnosis, psychotherapy, or a complementary therapy.
  Sophrology uses techniques such as: hypnosis, visualization, meditation, mindfulness, breathing exercises, gentle movements, body awareness...
  Sophrology techniques may be useful during medical procedures that cause stress and discomfort.
  Sophrology techniques may be useful during medical procedures that cause stress and discomfort.
  Patients will receive 6 sessions of sophrology
  Arms: Experimental arm : Speech therapy + Sophrology
Behavioral: Speech therapy — Speech therapy is a treatment that can help improve communication skills. patients will benefit from two speech therapy sessions per week for 6 months, lasting from 30 minutes to 1 hour depending on the patient's general condition.

SUMMARY:
Patients with brain tumours experience a loss of independence, which may occur suddenly or gradually. Communication with the patient may be rapidly impaired, due to impaired alertness, language and/or neurocognitive disorders.

In addition to these clinical symptoms, there is a high level of anxiety and depression in this population due to the severity of the diagnosis, with a major impact on the patients' quality of life. In this study, we are mainly interested in the proportion of this population with communication disorders where speech therapy is important In order to better take into account anxiety, which is often difficult to verbalise due to communication problems, sophrology can be proposed as an alternative to psychological support, which is often too complicated or inappropriate.

After having noted positive feedback from patients after joint speech therapy and sophrology treatment, we wish to evaluate the interest of coupling sophrology treatment for patients with glial tumours requiring speech therapy.

Our hypothesis is that this association would improve the level of anxiety, the quality of life and have a positive impact on the patient's speech therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven grade III and IV glial tumours requiring speech therapy;
* Patient willing to start outpatient speech therapy;
* Patient aged 18 years and over;
* Informed patient who has signed consent;
* Patient affiliated to a social security scheme.

Exclusion Criteria:

* Patient who has already had an initiation to sophrology in the context of his pathology;
* PS ≥ 4 ;
* Patients suffering from psychiatric disorders; delusional phases, schizophrenia against the practice of sophrology;
* Patient unable to follow the protocol (filling in questionnaires, attendance of sophrology and/or speech therapy sessions) for geographical, social or psychological reasons;
* Patients who do not speak French;
* Persons deprived of their liberty, under court protection, under curators or under the authority of a guardian.
* Women who are pregnant, likely to be pregnant or breastfeeding;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
The main objective is to compare the level of anxiety in the experimental arm with the control arm at 6 months. | 6 months
  Anxiety levels will be measured using the Hospital Anxiety and Depression Scale at 6 months in both treatment arms. The quality of life scale consists of 14 items scored from 0 to 3. A score of 0 indicates that the patient has no anxiety disorder, a score of 21 indicates that the patient has a severe anxiety disorder.

SECONDARY OUTCOMES:
The secondary objective is to evaluate the impact of the practice of sophrology on the patient's quality of life | 6 months
  Quality of life will be assessed by quality of life questionnaires at baseline and after 3 and 6 months of treatment. These are the QLQ-C30 v3 questionnaire and the brain-specific module EORTC-BN20 ;

CONTACTS AND LOCATIONS:
Overall Officials: CELINE THOMAS, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (1):
- Institut de Cancérologie de l'Ouest, Saint-Herblain, France